CLINICAL TRIAL: NCT00133419
Title: The Effect of Prophylactic Micronutrient Supplementation of Morbidity and Growth in HIV-infected and HIV-uninfected Children in South Africa
Brief Title: Micronutrients and Enteric Infections in African Children
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 00-095; NCT00156832 (obsolete NCT alias)
Record Dates: First submitted 2005-08-19; First posted 2005-08-23 (Estimated); Last update posted 2010-08-27 (Estimated); Status verified 2007-03

CONDITIONS: Enteric Infections
Keywords: micronutrient, supplementation, Africa, children, HIV
MeSH Terms: interventions — Vitamins; Zinc; Vitamin A

INTERVENTIONS:
Drug: Vitamin + Zinc + micronutrient mixture
Drug: Vitamin A
Drug: Vitamin A + Zinc

SUMMARY:
The purpose of the study is to see if giving vitamin and mineral supplements helps to protect infants and children from diarrhea, which vitamins and minerals help to improve a child's weight and growth, and if the same results occur in infants and children with HIV. HIV is the virus that causes AIDS. Study participants will include 516 infants aged 4-6 months. Participants will include: (1) HIV-infected children, (2) HIV-uninfected children with HIV-infected mothers, and (3) HIV-uninfected children with HIV-uninfected mothers. Subjects will have an equal chance of receiving one of three different vitamin and/or mineral supplements during the study. Study procedures will include up to 7 blood samples and stool samples every 3 months and body composition every 6 months. Participants will be involved in the study for up to 18 months.

DETAILED DESCRIPTION:
A major initiative to reduce the impact of enteric infections on health and nutrition has been micronutrient supplementation. Measures for routine vitamin A and zinc supplementation are gaining increasing support from international agencies, including UNICEF and the WHO. The primary objective of this study is to compare the effect of 3 micronutrient supplements (vitamin A only, vitamin A and zinc, and a micronutrient mixture containing vitamins A, B, C, D, E, K, and calcium, copper, folate, iodine, iron, magnesium and zinc) on prevalent days of diarrhea in 3 groups of children (HIV-infected children, HIV-uninfected children born to HIV-infected women, and HIV-uninfected children born to women without HIV infection). The secondary objectives of the study are: (1) to describe the pathogen-specific pattern of enteric infections in both HIV-infected and uninfected children during ages 6-24 months, with a focus on infection with C. parvum and other protozoan pathogens and (2) to conduct a cost-effectiveness analysis of micronutrient supplementation in children aged 6-24 months. The tertiary objectives of the study are: (1) to assess whether either zinc alone or a micronutrient mixture containing zinc affects linear growth and body composition and (2) to determine if infection with specific enteric pathogens is associated with the development of persistent diarrhea lasting > 14 days. The proposed study will be conducted through the African Centre for Health and Population Studies located in Hlabisa Health District, in northern KwaZulu Natal (KZN), South Africa. The study is a randomized, double blind, clinical controlled trial with 3 arms in a study population of infants stratified by HIV status and the HIV status of their mothers. Study participants will include a total of 516 infants aged 4-6 months. The following evaluations will be made throughout the study: (1) blood samples, (2) stool sampling-routine (collected at 6, 12, 18, and 24 months of age), (3) stool sampling-during diarrheal episodes, and (3) lean body mass and anthropometry (assessed at 6, 12, 18, and 24 months of age). Study participants will be involved in study related procedures for up to 18 months.

ELIGIBILITY:
Inclusion Criteria:

4-6 months of age (stratified by HIV status) Infant able to take oral preparations Consent of parent/guardian HIV status obtained from mother and child

Exclusion Criteria:

Documented micronutrient supplementation other than vitamin A in the preceding month Less than 60% of mean weight for age by NCHS guidelines (micronutrient intervention obligatory according to WHO guidelines for management of severely malnourished children) Persistent diarrhea (>=7 days) at the time of study enrollment Exclusive breastfeeding Infants in whom a second confirmatory HIV test cannot be obtained (when required) Co-enrollment of the infant in other clinical intervention trials e.g. antibiotic or vaccine trials

Ages: 4 Months to 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 516
Dates: Study Completion 2006-01

CONTACTS AND LOCATIONS:
Locations (1):
- Africa Centre for Health and Population Studies, Mtubatuba, South Africa

REFERENCES:
- [Derived] Chhagan MK, Van den Broeck J, Luabeya KK, Mpontshane N, Tomkins A, Bennish ML. Effect on longitudinal growth and anemia of zinc or multiple micronutrients added to vitamin A: a randomized controlled trial in children aged 6-24 months. BMC Public Health. 2010 Mar 18;10:145. doi: 10.1186/1471-2458-10-145. PMID 20298571
- [Derived] Chhagan MK, Van den Broeck J, Luabeya KK, Mpontshane N, Tucker KL, Bennish ML. Effect of micronutrient supplementation on diarrhoeal disease among stunted children in rural South Africa. Eur J Clin Nutr. 2009 Jul;63(7):850-7. doi: 10.1038/ejcn.2008.78. Epub 2009 Jan 28. PMID 19174830
- [Derived] Luabeya KK, Mpontshane N, Mackay M, Ward H, Elson I, Chhagan M, Tomkins A, Van den Broeck J, Bennish ML. Zinc or multiple micronutrient supplementation to reduce diarrhea and respiratory disease in South African children: a randomized controlled trial. PLoS One. 2007 Jun 27;2(6):e541. doi: 10.1371/journal.pone.0000541. PMID 17593956